CLINICAL TRIAL: NCT05087238
Title: Cognitive Behavior Therapy for Patients With Premature Ventricular Contractions - a Pilot Study
Brief Title: CBT for Premature Ventricular Contractions
Acronym: PVC-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Frieder Braunschweig, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVC-CBT
Record Dates: First submitted 2021-06-24; First posted 2021-10-21 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Premature Complexes
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVC-specific CBT (Other): This novel CBT treatment for symptomatic PVC targets cardiac anxiety and symptom preoccupation related to PVC. Treatment is developed from the research groups treatment for Atrial Fibrillation and may be altered during the treatment period to better meet the needs of the patients. Patients receive 10 weeks of CBT delivered through face to face digital video sessions.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — Cognitive Behavior Therapy for PVC-specific anxiety education, in-vivo exposure, interoceptive exposure, behavioral activation, relapse prevention

SUMMARY:
The purpose of the present interdisciplinary research program is to develop and evaluate a disease-specific cognitive behavior therapy (CBT) protocol to increase quality of life (QoL) and reduce symptom burden in patients with Premature Ventricular Contractions (PVC).

DETAILED DESCRIPTION:
Patients will be recruited in collaboration with arrythmia specialist units in Stockholm and through advertisement in local newspapers and social media. All patients giving informed consent will be screened thoroughly by the research nurse and a psychologist before included by the study cardiologist. 20-30 patients that meet eligibility criteria will be included and receive 8-10 sessions of cognitive behavior therapy during 8-10 weeks. Due to the current Covid-19 pandemic, treatment will be delivered face-to face through a secure digital platform. The psychologist delivering the treatment will have direct access to the study cardiologist during treatment. Follow-up at 3 and 6 months.

ELIGIBILITY:
Inclusion

* 18-70 years old
* PVCs that cause moderate to severe symptoms and leads to significant distress or interferes with daily life.
* Optimal medical treatment in the opinion of the treating physician.
* Able to read and write in Swedish.

Exclusion

* Structural heart disease including previous myocardial infarction, heart failure with preserved or reduced left ventricular ejection fraction, valvular disease, previous cardiac surgery.
* Other arrhythmia or severe medical illness;
* Scheduled for ablation therapy or any other cardiovascular intervention
* Any medical restriction to physical exercise.
* Severe depression or risk of suicide;
* Alcohol dependency.

All patients will undergo thorough cardiological and psychological assessment to ensure that eligibility criteria are met.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Premature Ventricular Contractions effect on Quality-of-life (PVCEQT) | baseline
  Version of the Atrial Fibrillation effects on Quality-of-life (AFEQT), adjusted to Premature Ventricular Contractions. Measures PVC-specific Quality of life in several domains. 14 questions graded on a 7 points likert scale. The total score ranges between 0 (severe symptoms and disability) and 98 (no symptoms and disability)
Premature Ventricular Contractions effect on Quality-of-life (PVCEQT) | 10 weeks from baseline
  Version of the Atrial Fibrillation effects on Quality-of-life (AFEQT), adjusted to Premature Ventricular Contractions. Measures PVC-specific Quality of life in several domains. 14 questions graded on a 7 points likert scale. The total score ranges between 0 (severe symptoms and disability) and 98 (no symptoms and disability)
Premature Ventricular Contractions effect on Quality-of-life (PVCEQT) | 5 months from baseline
  Version of the Atrial Fibrillation effects on Quality-of-life (AFEQT), adjusted to Premature Ventricular Contractions. Measures PVC-specific Quality of life in several domains. 14 questions graded on a 7 points likert scale. The total score ranges between 0 (severe symptoms and disability) and 98 (no symptoms and disability)
Premature Ventricular Contractions effect on Quality-of-life (PVCEQT) | 8 months from baseline
  Version of the Atrial Fibrillation effects on Quality-of-life (AFEQT), adjusted to Premature Ventricular Contractions. Measures PVC-specific Quality of life in several domains. 14 questions graded on a 7 points likert scale. The total score ranges between 0 (severe symptoms and disability) and 98 (no symptoms and disability)

SECONDARY OUTCOMES:
12-Item Short-Form Health Survey (SF-12) | baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 10 weeks from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 5 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 8 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
Symptom Checklist (SCL) | baseline
  Measures frequency and severity of 16 symptoms often experienced by patients with Atrial Fibrillation. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms. For total score sub scores are summed
Symptom Checklist (SCL) | 10 weeks from baseline
  Measures frequency and severity of 16 symptoms often experienced by patients with Atrial Fibrillation. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms. For total score sub scores are summed
Symptom Checklist (SCL) | 5 months from baseline
  Measures frequency and severity of 16 symptoms often experienced by patients with Atrial Fibrillation. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms. For total score sub scores are summed
Symptom Checklist (SCL) | 8 months from baseline
  Measures frequency and severity of 16 symptoms often experienced by patients with Atrial Fibrillation. Scoring range from 0 to 64 for frequency with a greater score indicating more frequent symptoms, and from range from 0 to 48 for severity, with a greater score indicating more severe symptoms. For total score sub scores are summed
Arrhythmia burden | baseline
  Number of premature ventricular contractions per 24 hours is assessed by 5-day ECG Holter-monitoring
Arrhythmia burden | 10 weeks from baseline
  Number of premature ventricular contractions per 24 hours is assessed by 5-day ECG Holter-monitoring
Arrhythmia burden | 8 months from baseline
  Number of premature ventricular contractions per 24 hours is assessed by 5-day ECG Holter-monitoring
Cardiac anxiety questionnaire (CAQ) | baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire (CAQ) | 10 weeks from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire (CAQ) | 5 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire (CAQ) | 8 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.

OTHER OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | baseline
  The PHQ-9 (26) is a well-established measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Patient Health Questionnaire-9 (PHQ-9) | 10 weeks from baseline
  The PHQ-9 (26) is a well-established measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Patient Health Questionnaire-9 (PHQ-9) | 5 months from baseline
  The PHQ-9 is a well-established measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Patient Health Questionnaire-9 (PHQ-9) | 8 months from baseline
  The PHQ-9 is a well-established measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Generalized Anxiety Disorder 7-item (GAD-7) | baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item (GAD-7) | 10 weeks from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item (GAD-7) | 5 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item (GAD-7) | 8 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Godin Shepard Leisure-time Physical Activity Questionnaire (GSLTPAQ) | baseline
  Measures level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numbers are the categorized in to low, moderate, and high levels of physical activity.
  measures changes in physical activity.
Godin Shepard Leisure-time Physical Activity Questionnaire (GSLTPAQ) | 10 weeks from baseline
  Measures level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numbers are the categorized in to low, moderate, and high levels of physical activity.
  measures changes in physical activity.
Godin Shepard Leisure-time Physical Activity Questionnaire (GSLTPAQ) | 5 months from baseline
  Measures level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numbers are the categorized in to low, moderate, and high levels of physical activity.
  measures changes in physical activity.
Godin Shepard Leisure-time Physical Activity Questionnaire (GSLTPAQ) | 8 months from baseline
  Measures level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numbers are the categorized in to low, moderate, and high levels of physical activity.
  measures changes in physical activity.
Body Sensation Questionnaire (BSQ) | baseline
  Measures fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire (BSQ) | 10 weeks from baseline
  Measures fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire (BSQ) | 5 months from baseline
  Measures fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire (BSQ) | 8 months from baseline
  Measures fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Client satisfaction Questionnaire (CSQ) | 10 weeks from baseline
  Measures treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
The Perceived stress scale (PSS-10) | baseline
  Measures levels of perceived stress, score ranging from 0 to 40, with a higher score indicating higher levels of experienced stress,
The Perceived stress scale (PSS-10) | 10 weeks from baseline
  Measures levels of perceived stress, score ranging from 0 to 40, with a higher score indicating higher levels of experienced stress,
The Perceived stress scale (PSS-10) | 5 months from baseline
  Measures levels of perceived stress, score ranging from 0 to 40, with a higher score indicating higher levels of experienced stress,
The Perceived stress scale (PSS-10) | 8 months from baseline
  Measures levels of perceived stress, score ranging from 0 to 40, with a higher score indicating higher levels of experienced stress,
Treatment Credibility Scale (TCS) | Will be measured 2 weeks from baseline
  Measures treatment credibility, scoring ranging between 0-50, with a higher score indicating higher levels of positive treatment expectations.
Adverse events | 10 weeks from baseline
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').

CONTACTS AND LOCATIONS:
Overall Officials: Frieder Braunschweig, Principal Investigator — Karolinska
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Liliequist BE, Sarnholm J, Skuladottir H, Olafsdottir E, Ljotsson B, Braunschweig F. Cognitive Behavioral Therapy for Symptom Preoccupation Among Patients With Premature Ventricular Contractions: Nonrandomized Pretest-Posttest Study. JMIR Cardio. 2024 May 7;8:e53815. doi: 10.2196/53815. PMID 38713500